CLINICAL TRIAL: NCT00301236
Title: A 5-Week Treatment, Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Fixed-Dose Study of the Efficacy, Tolerability and Safety of Dexmethylphenidate HCl Extended-Release Capsules Administered Once Daily in Pediatric Children With Attention-Deficit/Hyperactivity Disorder
Brief Title: Efficacy, Tolerability and Safety of Dexmethylphenidate HCl Extended-Release Capsules in Children With Attention-Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRIT124E2305
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: ADHD, ADD
Keywords: ADHD, children, CADS-T, Dexmethylphenidate-HCl, extended release
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

INTERVENTIONS:
Drug: Dexmethylphenidate HCl extended-release capsules

SUMMARY:
The purpose of this study is to determine which dosages of dexmethylphenidate HCl extended-release capsules may represent effective treatment for ADHD in children 6-12 years of age.

DETAILED DESCRIPTION:
The purpose of this study is to determine which dosages of dexmethylphenidate HCl extended-release capsules may represent effective treatment for ADHD in children 6-12 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 - 12 with a diagnosis of ADHD of any type , Same teacher who is willing to complete the assessment during the school term

Exclusion Criteria:

* Previous cardiac problems of the patient or the parents or current cardiac findings of the patient; Relevant medical condition other than ADHD; ADHD medication within a specified timeperiod prior to study start; Pregnancy or nursing; Positive drug screen

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 12 Years | Sex: All
Age Groups: Child
Enrollment: 252
Dates: Start 2006-02; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Assessment of the symptoms by the patient's teacher after 5 weeks of treatment.

SECONDARY OUTCOMES:
Assessment of the symptoms by the patient's parent after five weeks of treatment.
Change in severity of the illness assessed by the physician after 5 weeks of treatment
Improvement of the illness assessed by the physician after 5 weeks of treatment
Safety and tolerability of 5 week's treatment with dexmethylphenidate HCl extended-release capsules in children with Attention-Deficit/Hyperactivity Disorder by assessing the frequency of adverse findings

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (24):
- United States (24):
  - Novartis Investigational Site, Mesa, Arizona
  - Novartis Investigational Site, Little Rock, Arkansas
  - Novartis Investigational Site, Los Angeles, California
  - Novartis Investigational Site, Boulder, Colorado
  - Novartis Investigational Site, Maitland, Florida
  - Novartis Investigational Site, Orlando, Florida
  - Novartis Investigational Site, Stone Mountain, Georgia
  - Novartis Investigational Site, Libertyville, Illinois
  - Novartis Investigational Site, Overland Park, Kansas
  - Novartis Investigational Site, Prairie Village, Kansas
  - Novartis Investigational Site, Cambridge, Massachusetts
  - Novartis Investigational Site, Las Vegas, Nevada
  - Novartis Investigational Site, Piscataway, New Jersey
  - Novartis Investigational Site, Toms River, New Jersey
  - Novartis Investigational Site, New York, New York
  - Novartis Investigational Site, Staten Island, New York
  - Novartis Investigational Site, Chapel Hill, North Carolina
  - Novartis Investigational Site, Raleigh, North Carolina
  - Novartis Investigational Site, Columbus, Ohio
  - Novartis Investigational Site, Gresham, Oregon
  - Novartis Investigational Site, Philadelphia, Pennsylvania
  - Novartis Investigational Site, Jackson, Tennessee
  - Novartis Investigational Site, Memphis, Tennessee
  - Novartis Investigational Site, Houston, Texas